CLINICAL TRIAL: NCT04335045
Title: A Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PH100 Capsules in Healthy Adult Volunteers
Brief Title: Phase I Study of PH100 (Ecklonia Cava Phlorotannins)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phloronol Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-01-01
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Safety Issues
Keywords: Safety; Tolerability; Pharmacokinetics; PH100; Ecklonia cava; Phlorotannin

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, placebo-controlled, single ascending dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- 100mg Dose (Active Comparator): 1 x 100 mg PH100 capsule (n=6)
  Interventions: Drug: PH100 100mg
- Control for 100mg Dose (Placebo Comparator): 1 placebo capsule (n=2)
  Interventions: Drug: Placebo
- 200mg Dose (Active Comparator): 1 x 200 mg PH100 capsule (n=6)
  Interventions: Drug: PH100 200mg
- Control for 200mg Dose (Placebo Comparator): 1 placebo capsule (n=2)
  Interventions: Drug: Placebo
- 400mg Dose (Active Comparator): 2 x 200 mg PH100 capsules (n=6)
  Interventions: Drug: PH100 400mg
- Control for 400mg Dose (Placebo Comparator): 2 placebo capsules (n=2)
  Interventions: Drug: Placebo
- 800mg Dose (Active Comparator): 4 x 200 mg PH100 capsules (n=6)
  Interventions: Drug: PH100 800mg
- Control for 800mg Dose (Placebo Comparator): 4 placebo capsules (n=2)
  Interventions: Drug: Placebo
- 1200mg Dose (Active Comparator): 6 x 200 mg PH100 capsules (n=6)
  Interventions: Drug: PH100 1200mg
- Control for 1200mg Dose (Placebo Comparator): 6 placebo capsules (n=2)
  Interventions: Drug: Placebo
- 1600mg Dose (Active Comparator): 8 x 200 mg PH100 capsules (n=6)
  Interventions: Drug: PH100 1600mg
- Control for 1600mg Dose (Placebo Comparator): 8 placebo capsules (n=2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 1~8 Placebo capsule(s) corresponding to each PH100 dose
  Arms: Control for 100mg Dose; Control for 1200mg Dose; Control for 1600mg Dose; Control for 200mg Dose; Control for 400mg Dose; Control for 800mg Dose
Drug: PH100 100mg — 1 x 100 mg PH100 oral capsule
  Arms: 100mg Dose
Drug: PH100 200mg — 1 x 200 mg PH100 oral capsule
  Arms: 200mg Dose
Drug: PH100 400mg — 2 x 200 mg PH100 oral capsules
  Arms: 400mg Dose
Drug: PH100 800mg — 4 x 200 mg PH100 oral capsules
  Arms: 800mg Dose
Drug: PH100 1200mg — 6 x 200 mg PH100 oral capsules
  Arms: 1200mg Dose
Drug: PH100 1600mg — 8 x 200 mg PH100 oral capsules
  Arms: 1600mg Dose

SUMMARY:
The purpose of this study was to determine the safety and tolerability of PH100, a purified phlorotannins from a brown alga Ecklonia cava and the pharmacokinetics of its major compounds 8,8'-bieckol, dieckol, and phlorofucofuroeckol A (PFF-A), after single, ascending, oral doses of PH100 Capsules (over-encapsulated tablets) in healthy adult volunteers.

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, placebo-controlled, single ascending dose study in healthy volunteers in which subjects received either placebo or a 100 mg, 200 mg, 400 mg, 800 mg, 1200 mg, or 1600 mg dose of PH100 capsules (over-encapsulated tablets containing purified Ecklonia cava phlorotannins as an active ingredient) in escalating dose groups (six cohorts). A total of 48 subjects were enrolled. Each cohort comprised eight subjects. Within each cohort, six subjects received PH100 and two subjects received placebo. The first cohort was dosed as a single group with PH100 (100 mg) or placebo. The subsequent five cohorts were dosed sequentially with 200 mg, 400 mg, 800 mg, 1200 mg, and 1600 mg of PH100 or placebo. Safety and pharmacokinetic data were collected and evaluated following each cohort. Dose escalation occurred after review of the safety and pharmacokinetic data from the preceding cohort(s). Doses were administered with subjects in the fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant, nonbreastfeeding female;
* Between 40 and 75 years of age (inclusive);
* Body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and minimum weight of 50 kg (110 lbs);
* If female, subject was considered postmenopausal or surgically sterile and had status confirmed by one of the following:
* Physiologicallypostmenopausalbasedonnomensesforatleast2years(not due to lactational amenorrhea) and follicle stimulating hormone (FSH) levels equal to or greater than 40.0 mIU/mL at screening; or
* Bilateraloophorectomy,hysterectomy,orbilateraltuballigation(post 6 months). Or
* If female and of childbearing potential, subject agreed to use one of the following forms of birth control from 3 months prior through 12 days after study drug administration:
* Vasectomizedpartner(atleast6monthspriortodosing);
* Doublebarrier(diaphragmwithspermicide;condomswithspermicide);
* Intrauterinedevice(IUD);
* Abstinence(agreedtouseadoublebarriermethodiftheybecamesexually active during the study);
* Implantedorintrauterinehormonalcontraceptives;or
* Oral,patch,orinjectedcontraceptives,orvaginalhormonaldevice (i.e. NuvaRing®).
* If male, subject had a documented vasectomy or agreed to use a double-barrier local contraception (i.e., condom with spermicide) when engaging in sexual activity with women of childbearing potential from prior to the first dose of study drug through 28 days after the last dose of study drug;
* If male, subject agreed to refrain from sperm donation from prior to the first dose of study drug through 28 days after the last dose of study drug;
* Voluntarily consented to participate in this study and provided their written informed consent prior to start of any study-specific procedures;
* Able to communicate with the Investigator, and understand and comply with the requirements of the protocol;
* Willing and able to remain in the study unit for the entire duration of the confinement period and return for an outpatient visit;
* Had screening blood pressure (measured sitting after 3 minutes rest) 140/90 mmHg. Out-of-range blood pressure could be repeated once; and
* Willing and able to swallow up to eight size AAA capsules with water at dose administration. Size AAA capsules are 0.642 inches (16.31 mm) in length and 0.450 inches (11.44 mm) in diameter).

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, GI, endocrine (including thyroid), immunologic, dermatologic, neurologic, oncologic, respiratory, lymphatic, musculoskeletal, genitourinary, infective, inflammatory, connective tissue, or psychiatric disease or disorder or any other condition that, in the opinion of the Investigator, would have jeopardized the safety of the subject or the validity of the study results;
* Clinically relevant history or presence of cardiac arrhythmia, narrow angle glaucoma, benign prostatic hypertrophy (men only), Hashimoto's thyroiditis, lymphocytic thyroiditis, or uncontrolled diabetes;
* Had a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening;
* History or presence of allergic or adverse response to PH100 (product names: Seapolynol, Fibroboost, Fibronol, Seanol Longevity Plus, Circulate, Alginol, PC Ecklonia Cava, Seanol, Seanol-F, Seanol-EX, Seanol-TX, Venusen, Memories with Seanol-P, Astaxanthol, Brilliant Vision with Seanol-P, Gly-Control, Gyne-Andro-Plex, Lipid Balance, Seanol with Broccoraphanin, and Marine D3) or related drugs;
* Had used PH100 (product names: Seapolynol, Fibroboost, Fibronol, Seanol Longevity Plus, Circulate, Alginol, PC Ecklonia Cava, Seanol, Seanol-F, Seanol-EX, Seanol-TX, Venusen, Memories with Seanol-P, Astaxanthol, Brilliant Vision with Seanol-P, Gly-Control, Gyne-Andro-Plex, Lipid Balance, Seanol with Broccoraphanin, and Marine D3) as a supplement within 30 days prior to the first dose of study medication;
* Had been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication;
* Had donated blood or plasma within 30 days prior to the first dose of study medication;
* Had participated in another clinical trial (randomized subjects only) within 30 days prior to first dose of study medication;
* Had used any over-the-counter (OTC) medication, including nutritional supplements, within 5 half-lives or 14 days (whichever was longer) prior to the first dose of study medication;
* Had used any prescription medication, except hormonal contraceptives for women of childbearing potential or hormone replacement therapy, within 5 half-lives or 14 days (whichever was longer) prior to the first dose of study medication;
* Had ingested drinks or foods containing grapefruit or St. John's Wort within 14 days prior to the first dose of study medication;
* Had been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may have impacted subject safety or the validity of the study results;
* Had discontinued the use of implanted, intrauterine, or injected hormonal contraceptives less than 6 months prior to the first dose of study medication;
* Had discontinued the use of oral, patch, or vaginal hormonal contraceptives less than 1 month prior to the first dose of study medication;
* Had smoked or used tobacco products within 6 months prior to the first dose of study medication;
* Had a history of substance abuse or treatment (including alcohol);
* Was a female who had a positive pregnancy test result or was nursing, lactating, or trying to become pregnant;
* Had a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates), alcohol, or cotinine;
* Had a positive test for hepatitis B surface antigen (HbSAg), hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or had been previously treated for hepatitis B, hepatitis C, or HIV infection; or
* Had difficulty swallowing up to eight capsules.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2014-12-08 (Actual); Study Completion 2014-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 96 hours postdose
  Subjects were instructed to inform the study physician and/or research personnel of any AEs that occurred at any time during the study. Subjects were monitored for AEs from the beginning of confinement through the end-of-study visit (96 hours after dose administration). Reported or observed AEs were documented and followed to resolution.
Hematocrit (%) | 48 hours postdose
  Safety Assessment in Hematology
Hemoglobin (g/dL) | 48 hours postdose
  Safety Assessment in Hematology
Erythrocytes (10^6/uL) | 48 hours postdose
  Safety Assessment in Hematology
Leukocytes (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Basophils (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Basophils/Leukocytes (%) | 48 hours postdose
  Safety Assessment in Hematology
Eosinophils (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Eosinophils/Leukocytes (%) | 48 hours postdose
  Safety Assessment in Hematology
Lymphocytes (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Lymphocytes/Leukocytes (%) | 48 hours postdose
  Safety Assessment in Hematology
Monocytes (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Monocytes/Leukocytes (%) | 48 hours postdose
  Safety Assessment in Hematology
Neutrophils (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Neutrophils/Leukocytes (%) | 48 hours postdose
  Safety Assessment in Hematology
Platelets (10^3/uL) | 48 hours postdose
  Safety Assessment in Hematology
Serum Glucose (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Sodium (mmol/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Potassium (mmol/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Calcium (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Chloride (mmol/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Blood urea nitrogen (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Creatinine (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Urate (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Albumin (g/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Alkaline phosphatase (U/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Aspartate phosphatase (U/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Alanine transaminase (U/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Total bilirubin (mg/dL) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Lactate Dehydrogenase (U/L) | 48 hours postdose
  Safety Assessment in Serum Chemistry
Specific gravity | 48 hours postdose
  Safety Assessment in Urinalysis
pH | 48 hours postdose
  Safety Assessment in Urinalysis
Glucose (mg/dL) | 48 hours postdose
  Safety Assessment in Urinalysis
Nitrite (Negative/Positive) | 48 hours postdose
  Safety Assessment in Urinalysis
Leukocyte esterase (/uL) | 48 hours postdose
  Safety Assessment in Urinalysis
Occult blood (/uL) | 48 hours postdose
  Safety Assessment in Urinalysis
Bilirubin (mg/dL) | 48 hours postdose
  Safety Assessment in Urinalysis
Urobilinogen (mg/dL) | 48 hours postdose
  Safety Assessment in Urinalysis
Change from Baseline Systolic Blood Pressure (mmHg) | 2, 4, 48, 96 hours postdose
  Safety Assessment in Vital Signs
Change from Baseline Diastolic Blood Pressure (mmHg) | 2, 4, 48, 96 hours postdose
  Safety Assessment in Vital Signs
Change from Baseline Pulse Rate (bpm) | 2, 4, 48, 96 hours postdose
  Safety Assessment in Vital Signs
Change from Baseline Respiration Rate (Breath/Min) | 2, 4, 48, 96 hours postdose
  Safety Assessment in Vital Signs
Change from Baseline Body Temperature (degrees C) | 2, 4, 48, 96 hours postdose
  Safety Assessment in Vital Signs
ECG heart rate (bpm) | 48 hours postdose
  Safety Assessment in ECG
PR interval (ms) | 48 hours postdose
  Safety Assessment in ECG
QRS complex (ms) | 48 hours postdose
  Safety Assessment in ECG
QT interval (ms) | 48 hours postdose
  Safety Assessment in ECG
QTcB interval (ms) | 48 hours postdose
  Safety Assessment in ECG
QTcF interval (ms) | 48 hours postdose
  Safety Assessment in ECG

SECONDARY OUTCOMES:
Change in Blood Concentration of 8,8'-bieckol (ng/mL) by HPLC-MS | at 0, 15, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 96 hours after dosing.
  Pharmacokinetics of 8,8'-bieckol, a major compound of PH100, after single, ascending, oral doses (100 mg, 200 mg, 400 mg, 800 mg, 1200 mg, and 1600 mg) of PH100 in normal healthy volunteers.
Change in Blood Concentration of dieckol (ng/mL) by HPLC-MS | at 0, 15, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 96 hours after dosing.
  Pharmacokinetics of 8,8'-bieckol, a major compound of PH100, after single, ascending, oral doses (100 mg, 200 mg, 400 mg, 800 mg, 1200 mg, and 1600 mg) of PH100 in normal healthy volunteers.
Change in Blood Concentration of PFF-A (ng/mL) by HPLC-MS | at 0, 15, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 96 hours after dosing.
  Pharmacokinetics of 8,8'-bieckol, a major compound of PH100, after single, ascending, oral doses (100 mg, 200 mg, 400 mg, 800 mg, 1200 mg, and 1600 mg) of PH100 in normal healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: George J. Atiee, MD, Principal Investigator — Worldwide Clinical Trials Early Phase Services, LLC
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No